CLINICAL TRIAL: NCT03836157
Title: Phase II Trial of Mirvetuximab Soravtansine (IMGN853) and Bevacizumab in Patients With Endometrial Cancer
Brief Title: Mirvetuximab Soravtansine (IMGN853) and Bevacizumab in Patients With Endometrial Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not initiated.
Sponsor: University of Oklahoma (Other)
Collaborators: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUSCC-IMGN-001
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Endometrial Cancer; Endometrial Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma
Keywords: Mirvetuximab soravtansine; gynecologic cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — mirvetuximab soravtansine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mirvetuximab and Bevacizumab (Experimental): * Mirvetuximab Soravtansine 6mg/kg IV (adjusted ideal body weight), on day 1 of each 21 day cycle.
  * Bevacizumab 15 mg/kg, IV, on day 1 of each 21-day cycle.
  Interventions: Drug: Mirvetuximab Soravtansine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine — The dose will not be recalculated unless the patient has ±10% weight change.
  Other Names: IMGN853
Drug: Bevacizumab — Subject will receive IMGN853 first followed by bevacizumab. There is no planned delay between the IMGN853 and bevacizumab administration.

SUMMARY:
IMGN853 is designed to inhibit cell division and cell growth of folate receptor 1 (FRα)-expressing tumor cells. The purpose of this study is to test the safety of IMGN853 and bevacizumab and see what effects (good and bad) that this combination treatment has on subjects with recurrent endometrial cancer.

DETAILED DESCRIPTION:
SCREENING: During the screening portion of the study, the subject will need to have tumor tissue tested and other exams to determine if s/he may proceed to the treatment part of the study. The subject's tumor tissue will be tested from either a previous or recent surgery or biopsy to see if it contains the FRα protein. If the tumor is positive and the patient meets all other eligibility, then the subject may proceed to treatment.

TREATMENT: Study drugs (IMGN853 and bevacizumab) will be given by vein (IV) once each cycle on day 1 of 21 day cycle.

Regular cancer care exams, tests, and procedures will occur. Additionally, an eye doctor visit with complete eye examination every other treatment cycle. Subjects will also self-administer eye drops as prescribed by the eye doctor.

Study participation is up to three years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological diagnosis of endometrial carcinoma (including others per protocol).
2. Expression of folate receptor alpha (FRα) on either archival tumor or new biopsy is required.
3. Measurable disease
4. Evidence that the endometrial cancer is advanced, recurrent, or persistent and has relapsed or is refractory to curative therapy or established treatments.
5. At least 1 prior platinum-based chemotherapeutic regimen, but not more than 2 prior chemotherapeutic regimens, for management of endometrial carcinoma. Prior treatment may include chemotherapy, or chemotherapy/radiation therapy . Chemotherapy administered in conjunction with primary radiation as a radio-sensitized therapy will be considered a systemic chemotherapy regimen
6. Female patients 18 years or older
7. Eastern Cooperative Oncology Group performance status of 0 to 1;
8. Patient must have archival tumor tissue available from the primary or recurrent cancer prior to first dose. If archival tumor sample is not available, tumor sample from new biopsy is acceptable.
9. Patients must have acceptable organ and marrow function as defined per protocol
10. Time from prior therapy:

    1. Systemic anti-neoplastic therapy: five half-lives or four weeks, whichever is shorter. Hormonal therapy is not considered anti-neoplastic therapy.
    2. Radiotherapy: wide-field radiotherapy (e.g. > 30% of marrow-bearing bones) completed at least four weeks, or focal radiation completed at least two weeks, prior to starting study treatment
11. Patients must have a life expectancy of at least 3 months
12. Patients should have no major existing co-morbidities or medical conditions that will preclude therapy
13. Ability to understand and the willingness to sign a written informed consent document, and to comply with the requirements of the protocol; with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
14. Female patients of reproductive potential and their male partners must agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through at least twelve weeks after the last dose of IMGN853 and/ or bevacizumab.

Exclusion Criteria:

1. Previous treatment with mirvetuximab.
2. Invasive cancer within the past 2 years. Noninvasive non-melanoma skin cancers are not exclusions if they have undergone complete resection.
3. Untreated or symptomatic central nervous system (CNS) metastases. Patients with asymptomatic CNS metastases are eligible provided they have been clinically stable for at least 4 weeks prior to first dose of study treatment), have no evidence of new or emerging CNS metastasis, and are not using steroids for at least 7 days prior to first dose of study treatment.
4. Unstable angina or myocardial infarction within the previous 6 months; uncontrolled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications); prior history of hypertensive crisis or hypertensive encephalopathy; symptomatic congestive heart failure (NYHA Class III and IV); uncontrolled cardiac arrhythmia; clinically-significant vascular disease (e.g. aortic aneurysm, or dissecting aneurysm), severe aortic stenosis; clinically significant peripheral vascular disease; history of any CNS cerebrovascular ischemia or stroke within the last 6 months.
5. Active pulmonary disease or other coexisting medical condition that would preclude full compliance with the study.
6. Receiving any other investigational agents.
7. History of prior severe infusion reaction to a monoclonal antibody. Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies.
8. Persisting ≥Grade 2 toxicity (except alopecia) from previous anti-cancer treatment.
9. Patients with > Grade 1 peripheral neuropathy
10. Active or chronic corneal disorder, including but not limited to the following:

    * Sjogren's syndrome
    * Fuchs corneal dystrophy (requiring treatment)
    * History of corneal transplantation
    * Active herpetic keratitis
    * Active ocular conditions requiring on-going treatment/monitoring such as wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, presence of papilledema, and monocular vision.
11. Serious concurrent illness or clinically-relevant active infection, including but not limited to the following:

    * Known active hepatitis B or C
    * Known Human Immunodeficiency Virus (HIV) infection
    * Varicella-zoster virus (shingles)
    * Cytomegalovirus infection
    * Any other known concurrent infectious disease, requiring IV antibiotics within 2 weeks of study enrollment
12. History of cirrhotic liver disease
13. History or evidence of thrombotic or hemorrhagic disorders within 6 months before first study treatment
14. Required used of folate-containing supplements (e.g. for folate deficiency)
15. Pregnancy
16. History of bowel obstruction (including subocclusive disease) related to underlying disease within 6 months of study treatment.
17. Clinically-significant proteinuria defined per protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-31 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Response rate of patients who remain progression free | 6 months
Percentage of patients who remain progression free | 6 months

SECONDARY OUTCOMES:
Incidence of adverse events | up to 3 years
Progression free survival | up to 3 years
Overall survival | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No